CLINICAL TRIAL: NCT03592368
Title: Neurocognitive Targets of Hostile Interpretation Bias Training to Treat Irritability
Brief Title: Hostile Interpretation Bias Training to Treat Irritability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-0464
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Irritable Mood; Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active IBT, Out of MRI (Active Comparator): Interpretation bias training where participants learn more positive judgements of ambiguous facial expressions relative to their own baseline bias. This arm is completed in the clinic.
  Interventions: Device: IBT
- Sham IBT, Out of MRI (Sham Comparator): Interpretation bias training where participants' baseline judgements of ambiguous facial expressions is reinforced. This arm is completed in the clinic.
  Interventions: Device: IBT
- Active IBT, In MRI (Active Comparator): Interpretation bias training where participants learn more positive judgements of ambiguous facial expressions relative to their own baseline judgments. This arm is completed in a magnetic resonance imaging machine.
  Interventions: Device: IBT
- Sham IBT, In MRI (Sham Comparator): Interpretation bias training where participants' baseline judgements of ambiguous facial expressions is reinforced. This arm is completed in a magnetic resonance imaging machine.
  Interventions: Device: IBT

INTERVENTIONS:
Device: IBT — Interpretation bias training

SUMMARY:
Hostile interpretation bias may be a feature of severe, chronic irritability in children, one of the most common psychiatric symptoms of childhood. Interpretation bias training (IBT) is a computer-based training program that may reduce irritability in youths. This trial lays the groundwork for a test IBT on irritability.

DETAILED DESCRIPTION:
This trial lays the foundation for a preliminary test of efficacy of IBT on irritability by establishing IBT's neurocognitive treatment targets: hostile interpretation bias and response in the neural threat-learning system.

The design is a single-blinded, randomized controlled trial of IBT on its targets. The study will have four arms, with 25 participants in each arm for all four conditions of training (active versus sham) and scanning (in MRI or out of MRI scanner). During IBT, participants judge as happy or angry facial expressions which are on a continuum between happy and angry. The point at which judgments shift from predominantly happy to angry on this continuum is the indifference point. During training feedback encourages no change in the indifference point or a change in the indifference point towards more happy judgments of ambiguous faces. A shift in indifference point towards more benign judgments is interpreted as a reduction in hostile interpretation.

The design will test whether active relative to sham IBT shifts the indifference point towards more benign judgments. Neural response to active versus sham IBT will be measured in half the sample.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in mental health treatment, with at least:

  1. mild, clinically significant irritability, and
  2. typical intellectual functioning (IQ>80)

Exclusion Criteria:

* Any of the following mental health diagnoses:

  1. current post-traumatic stress
  2. lifetime bipolar I or II disorder
  3. lifetime cyclothymic disorder
  4. lifetime psychotic disorder
  5. lifetime autism spectrum disorder
* Major medical problems, including head trauma.
* MRI-specific safety exclusions for the MRI arms.
* Clinical instability.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stoddard, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
A commitment to data sharing and analytic code has been made. Specifics of the data sharing plan require further work due to the collection of protected health information.

REFERENCES:
- [Background] Stoddard J, Sharif-Askary B, Harkins EA, Frank HR, Brotman MA, Penton-Voak IS, Maoz K, Bar-Haim Y, Munafo M, Pine DS, Leibenluft E. An Open Pilot Study of Training Hostile Interpretation Bias to Treat Disruptive Mood Dysregulation Disorder. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):49-57. doi: 10.1089/cap.2015.0100. Epub 2016 Jan 8. PMID 26745832
- [Background] Haller SP, Stoddard J, Botz-Zapp C, Clayton M, MacGillivray C, Perhamus G, Stiles K, Kircanski K, Penton-Voak IS, Bar-Haim Y, Munafo M, Towbin KE, Brotman MA. A Randomized Controlled Trial of Computerized Interpretation Bias Training for Disruptive Mood Dysregulation Disorder: A Fast-Fail Study. J Am Acad Child Adolesc Psychiatry. 2022 Jan;61(1):37-45. doi: 10.1016/j.jaac.2021.05.022. Epub 2021 Jun 17. PMID 34147585
- [Background] Stoddard J, Haller SP, Costa V, Brotman MA, Jones M. A Computational Model Reveals Learning Dynamics During Interpretation Bias Training With Clinical Applications. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Oct;8(10):1033-1040. doi: 10.1016/j.bpsc.2023.03.013. Epub 2023 Apr 14. PMID 37062362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active IBT, Out of MRI | Sham IBT, Out of MRI | Active IBT, In MRI | Sham IBT, In MRI
Started | 29 | 26 | 20 | 22
Completed | 28 | 24 | 20 | 21
Not Completed | 1 | 2 | 0 | 1
Not completed — Per protocol, randomized but not exposed to intervention due to COVID policy | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Per protocol, received intervention but with inadequate engagement for arm inclusion | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active IBT, Out of MRI | Sham IBT, Out of MRI | Active IBT, In MRI | Sham IBT, In MRI | Total
Number analyzed (Participants) | 28 | 24 | 20 | 21 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.31) | 14.8 (1.45) | 15.2 (1.55) | 15.2 (1.27) | 15.1 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 11 | 11 | 54
  Male | 9 | 11 | 9 | 10 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 4 | 9
  Not Hispanic or Latino | 25 | 23 | 19 | 17 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 23 | 23 | 15 | 19 | 80
  More than one race | 3 | 1 | 3 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 20 | 21 | 93
Indifference Point [Mean (Standard Deviation); unit: units on a morph continuum scale] | 5.60 (1.40) | 5.49 (1.13) | 6.37 (6.50) | 5.29 (1.36) | 5.66 (1.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Interpretation Bias
Description: Interpretation bias is measured by the indifference point of happy-angry judgments of a continuum of 15 images of face emotion expression that are morphed between completely happy=1 to completely angry=15 facial expressions. Indifference point is represented on this scale of 1 to 15 faces. It represents the point on the face continuum where judgements change from predominantly happy to predominantly angry. Indifference points have a minimum value of 1 and a maximum value of 15, though are typically in the middle of the face-emotion continuum, e.g. 7. Lower indifference points represent a higher bias towards hostile (or angry) judgments. Change in interpretation bias is the difference between the post- and pre-training indifference points. This can range from -14 to 14, with positive numbers reflecting the degree to which the happy/angry decision bias is shifted towards more happy judgements. High positive numbers reflect a greater increase in happy judgments.
Time Frame: Up to one day before and after the single 1 day training session of Interpretation bias training session.
Population: Arms are collapsed across completing IBT in or out of the scanner.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active IBT; Sham IBT: IBT: Interpretation bias training
Arm/Group | Active IBT | Sham IBT
Number analyzed (Participants) | 48 | 45
units on a scale | 1.53 (1.05) | 0.55 (1.14)
Statistical Analysis 1: Comparison: Active IBT vs Sham IBT; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: Neural Response in Threat Learning System.
Description: Amygdala functional connectivity to ventromedial prefrontal cortex is measured by covariance in fluctuations in blood oxygen-level dependent signal between these regions during functional magnetic resonance imaging (fMRI) during the course of training. The outcome measure is a count of these randomized participants for whom the fMRI measure is valid for the planned connectivity analysis. These participants completed the task in scanner with acceptable behavioral data and fMRI data. Quality control for fMRI included visual inspection of brain images for quality, coverage, and proper alignment across functional, anatomic and template images. The fMRI images passed analysis benchmarks of <20% censored volumes and <0.25 mm Euclidean distance average censored motion across the task. Censor thresholds are 0.3 mm Euclidean distance and 5% voxels with outlying intensity values.
Time Frame: During the course of the 1 day single session of interpretation bias training session.
Measure: Count of Participants; unit: Participants
Arm/Group | Active IBT, In MRI | Sham IBT, In MRI
Number analyzed (Participants) | 20 | 22
Participants | 16 | 18

3. Secondary Outcome: Learning Rate
Description: Learning rate as measured by a reinforcement learning computational model during IBT, please see the reference Stoddard et al., 2023, for model details. As in general reinforcement learning models, it is the proportion of prediction error that is applied to future expectations. In this trial, when a participant received feedback about a judgement they made of a face, the participant implicitly compares that feedback to their expectations about that face. The difference between the feedback and their expectations is called prediction error. The learning rate the proportion of this prediction error that is applied to future expectations across the learning session. In that way it represents learning. Learning rate is a continuous, unitless value. It ranges from 0, representing no learning, to 1, representing perfect learning. It is generally small. The learning rate reported here is its form estimated across face emotions (see Stoddard et al., 2023).
Time Frame: During the course of the 1 day single interpretation bias training session.
Population: Collapsed across the in and out of scanner groups.
Measure: Median (Inter-Quartile Range); unit: proportion of prediction error
Arm/Group | Active IBT | Sham IBT
Number analyzed (Participants) | 48 | 45
proportion of prediction error | 0.019 [0.0098 to 0.039] | 0.017 [0.0082 to 0.032]
Statistical Analysis 1: Comparison: Active IBT vs Sham IBT; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Irritability
Description: Irritability is the tendency towards anger and temper outburst as measured by the Affective Reactivity Index, a seven item scale. Each item has 3 response options which are coded as follows: "not true"=0, "somewhat true"=1, and "certainly true"=2. The first six items are summed to generate a total score that reflects the degree over irritability over the past week. The Affective Reactivity Index ranges from 0 to 12. Higher values reflect more irritability. What is reported here is the average post- minus pre-treatment score, by parent report. In these differences, negative values are in the unit of this scale and the absolute value represents the degree of irritability reduction.
Time Frame: Within one week prior to Interpretation bias training and one week +/- 3 days after Interpretation bias training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active IBT | Sham IBT
Number analyzed (Participants) | 48 | 45
score on a scale | -2.04 (2.07) | -1.44 (2.65)
Statistical Analysis 1: Comparison: Active IBT vs Sham IBT; Test type: Superiority; p = 0.12, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between randomization and the intervention (up to one week) and through the follow up period following IBT (one week) after interpretation bias training.
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definition. Adverse event information was collected on follow up query for any clinically significant change.
Arm/Group | Active IBT, Out of MRI | Sham IBT, Out of MRI | Active IBT, In MRI | Sham IBT, In MRI
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26 | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/20 | 1/22
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 1/20 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active IBT, Out of MRI (N=29) | Sham IBT, Out of MRI (N=26) | Active IBT, In MRI (N=20) | Sham IBT, In MRI (N=22)
Suicidal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for aborted suicide attempt following family argument. Occurred after randomization but prior to exposure to intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active IBT, Out of MRI (N=29) | Sham IBT, Out of MRI (N=26) | Active IBT, In MRI (N=20) | Sham IBT, In MRI (N=22)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Expressed suicidal ideation in direct response to school stressor (with method and intent) but no plan or behavior. Emergency evaluation resulted in discharge to current outpatient care with no increase in level of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03592368/Prot_SAP_001.pdf
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03592368/ICF_000.pdf